CLINICAL TRIAL: NCT01780818
Title: A Randomized, Controlled Trial Comparing Air Insufflation, Water Immersion and Water Exchange During on Demand Sedation Colonoscopy in CRC Screening Patients
Brief Title: A Comparison of Air Insufflation, Water Immersion and Water Exchange Colonoscopy in CRC Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Presidio Ospedaliero Santa Barbara (Other)
Responsible Party: Principal Investigator, Sergio Cadoni, M.D., Responsabile Servizio Endoscopia Digestiva, Presidio Ospedaliero Santa Barbara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PG.2012.27110; ASL07_WW-2012 (Other: S. Barbara Hospital, Iglesias (CA), Italy)
Record Dates: First submitted 2013-01-28; First posted 2013-01-31 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Pain; Colorectal Adenomas; Colorectal Cancer
Keywords: Warm Water Infusion colonoscopy; Water Immersion colonoscopy; Water Exchange colonoscopy; Painless unsedated colonoscopy; Adenoma detection rate; Adenoma resection rate
MeSH Terms: conditions — Pain; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Air insufflation method. (Active Comparator): Colonoscopy will be performed in the standard fashion, with the minimal air insufflation required to aid insertion and allowing for washing as needed. Considered to be standard procedure.
  Interventions: Other: Air Insufflation method.
- Water Immersion method. (Experimental): Air will not be insufflated until the cecum is reached. It will be allowed only 3 times and no more than 10 seconds each time (ITT failure if >3) if the lumen cannot be seen. Infusion of water during the insertion phase of colonoscopy mainly to open the colonic lumen and progress to the cecum immersed in the water environment thus created, without attempting to clear the colon contents. Residual air in the colon will not be removed. Infused water and residual feces will be suctioned back predominantly during withdrawal.
  Interventions: Other: Water Immersion method.
- Water Exchange method. (Experimental): Air will not be insufflated until the cecum is reached. Infusion of a sufficient amount of water to render the lumen of the colon a slit to progress with the colonoscope. Part of the infused water will be constantly suctioned back exchanging clean for dirty or hazy water. Suction of water will also be applied when colonoscope insertion proceeds smoothly. Air pockets will be always aspirated to collapse the lumen. After cecal intubation as much residual water as possible will be aspirated before beginning the withdrawal phase. During withdrawal residual water and feces will be suctioned.
  Interventions: Other: Water Exchange method.

INTERVENTIONS:
Other: Air Insufflation method. — Colonoscopy will be performed in the standard fashion, with the minimal air insufflation required to aid insertion and allowing for washing as needed. Considered to be standard procedure.
  Arms: Air insufflation method.
Other: Water Immersion method. — Air will not be insufflated until the cecum is reached. It will be allowed only 3 times and no more than 10 seconds each time (ITT failure if >3) if the lumen cannot be seen. Infusion of water during the insertion phase of colonoscopy mainly to open the colonic lumen and progress to the cecum immersed in the water environment thus created, without attempting to clear the colon contents. Residual air in the colon will not be removed. Infused water and residual feces will be suctioned back predominantly during withdrawal.
  Arms: Water Immersion method.
Other: Water Exchange method. — Air will not be insufflated until the cecum is reached. Infusion of a sufficient amount of water to render the lumen of the colon a slit to progress with the colonoscope. Part of the infused water will be constantly suctioned back exchanging clean for dirty or hazy water. Suction of water will also be applied when colonoscope insertion proceeds smoothly. Air pockets will be always aspirated to collapse the lumen. After cecal intubation as much residual water as possible will be aspirated before beginning the withdrawal phase. During withdrawal residual water and feces will be suctioned.
  Arms: Water Exchange method.

SUMMARY:
Water-aided method for colonoscopy can be broadly subdivided into two major categories. Water Immersion (WI), characterized by suction removal of the infused water predominantly during the withdrawal phase of colonoscopy, and Water Exchange (WE), characterized by suction removal of infused water predominantly during the insertion phase of colonoscopy. Several studies showed that WE significantly reduces pain compared to WI and colonoscopy with traditional air insufflation (AI), increases the number of unsedated procedures and adenoma detection rate (ADR), in particular proximal ADR. This randomized controlled trial will be a direct comparison of Air Insufflation, Water Immersion and Water Exchange to test the hypothesis that WAC (particularly WE) would significantly decrease pain score during colonoscopy in average-risk screening patients. Several other secondary outcomes will also be analyzed.

DETAILED DESCRIPTION:
Introduction

Water-aided methods for colonoscopy can be broadly subdivided into two major categories. Water Immersion (WI) is characterized by suction removal of the infused water predominantly during the withdrawal phase of colonoscopy and Water Exchange (WE) is characterized by suction removal of infused water predominantly during the insertion phase of colonoscopy. Several studies showed that WE significantly reduces pain compared to WI and colonoscopy with traditional air insufflation (AI), increases the number of unsedated procedures and adenoma detection rate (ADR), in particular proximal ADR. This randomized controlled trial will be a direct comparison of Air Insufflation, Water Immersion and Water Exchange to test the hypothesis that WAC (particularly WE) would significantly decrease pain score during colonoscopy in average-risk screening patients. Several other secondary outcomes will also be analyzed.

Method

Examinations will be allocated to Water Exchange, Water Immersion or Air Insufflation during the insertion phase of colonoscopy based on a computer generated random list. Procedures will be started by 6 board-certified endoscopists, three with experience in 8,000-10,000 and three with experience in 2,000-5,000 colonoscopies with AI, 285 with WI and 890 with WE overall. High-resolution wide-angle variable-stiffness adult video colonoscopes (Olympus HD 180 series; Olympus Corp, Hamburg, Germany) will be used. Need to change to a smaller caliber colonoscope will be considered ITT failure.

Patients will have a low volume split dose bowel preparation with 2L of polyethylene glycol (PEG) solution or Sodium Picosulfate. Investigators will be blinded to the colon preparation used. Before starting the procedure, a questionnaire recording demographic data, previous abdominal surgery, co-morbidities and current medications will be administered by the endoscopists. The patients, but not endoscopists and assisting nurses, will be blinded to the method used. At discharge the patient will be asked to guess which method has been used. If no more than half of the responses are correct, patients' blinding will be considered adequate.

Colonoscopy will begin with the patients in the left lateral position, without premedication.

The withdrawal phase will be identical in all arms of the study using air insufflation to obtain adequate distension of the colonic lumen for mucosal inspection, biopsy and/or polypectomy.

Patients randomized to the water-aided colonoscopy group, during the insertion phase after reaching the rectosigmoid junction, will have the colon irrigated with water at 37°C maintained with a water bath. Infusions will be performed using flushing pumps (Olympus OFP2, Olympus, Hamburg, Germany or Velocity irrigation pump, US Endoscopy, OH, USA). There will be no restriction of the overall volume of water that can be infused to get adequate lumen distention and reach the cecum. With the patient in the left lateral position water infused into the colon at the rectal sigmoid junction flows into the descending colon. The weight of the water in the left side of the colon straightens the sigmoid segment increasing the ease of insertion and reducing the risk of loop formation. The air pump will be turned off to avoid inadvertent insufflation.

Water Immersion will involve the infusion of water during the insertion phase of colonoscopy mainly to open the colonic lumen and progress to the cecum immersed in the water environment thus created, without attempting to clear the colon contents. Use of water as an adjunct to air insufflation to facilitate insertion and removal of infused water predominantly during withdrawal are characteristic features of WI. This traditional adjunct facilitates passage through the sigmoid colon with severe diverticulosis, speeds arrival to the splenic flexure, decreases colonic spasm, minimizes pain, and even enhances cecal intubation in previously incomplete colonoscopies. Residual air in the colon will not be removed. The infused water and residual feces will be suctioned back only during withdrawal. Air insufflation will be allowed if the lumen cannot be seen and the endoscopists judges unsafe to advance the colonoscope. It will last no more than 10 seconds and will be recorded in the patient data sheet. If more than 3 episodes of air insufflation will be recorded the procedure will be considered ITT failure.

Water Exchange will involve complete exclusion of air insufflation, removal of residual colonic air and feces and of infused water predominantly during insertion to assist identification of the lumen. WE minimizes loop formation and decreases discomfort. By providing salvage cleansing during insertion, WE allows the colonoscopist to devote a greater proportion of the withdrawal to inspection. WE will involve the infusion of a sufficient amount of water to open the lumen of the colon to allow passage of the instrument, thus rendering the colonic lumen a slit to progress with the colonoscope. If the lumen does not open, the colonoscope will be slightly retracted and the infusion started again. Part of the infused water will be constantly suctioned back exchanging clean for dirty or hazy water. Suction of infused water will also be applied when colonoscope insertion proceeds smoothly. Air pockets, when encountered, will be always aspirated to collapse the lumen: the absence of air space forces the colonoscopist to use water to clear residual feces and to find the way through the colon. Removal of the air also shortens the colon and takes out all the sharp turns at the flexures and redundant segments, reducing the risk of loop formation: water instillation does not elongate the colon as much as air insufflation does. In a collapsed, airless colon turbulences created at the tip of the instrument facilitate the removal by suction of residual feces adherent to the mucosa. This provides salvage cleansing during the insertion phase. After cecal intubation as much residual water as possible will be aspirated before beginning the withdrawal phase. During withdrawal scarce amounts of water are left to aspirate, and residual water and feces will be suctioned.

In the AI group, colonoscopy will be performed in the standard fashion, allowing for washing as needed. In all groups abdominal compression and position change were applied as needed.

Cecal intubation will be defined as passage of the tip of the colonoscope to a point proximal to the ileocecal valve with adequate visualization of the cecum and appendix orifice. A stopwatch will be used to time the procedures. Cecal intubation time will be defined as the time for passage of the colonoscope from the rectum to the cecum. The withdrawal phase will last at least 6 minutes. Polyp resection will be done during withdrawal in all groups. Time for polypectomy or biopsy will add to the total colonoscopy time. Pathology reports of all polyps will be reviewed and recorded to evaluate adenoma detection rate (ADR, defined as the proportion of subjects with at least one adenoma of any size), the location, the total number of adenomas resected per subject (ARR), and the percentage of subjects with advanced adenomas. The amount of water infused during insertion and withdrawal, the number of position changes and any adverse outcome will be recorded. Cardiopulmonary function will be monitored. Significant oxygen desaturation (<85% for >15 seconds) will be recorded. Vagal reaction will be defined as heart rate <60 beats per minute accompanied by excessive sweating, nausea and/or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive 50 to 70 year-old first time average-risk screening patients agreeing to start procedure without premedication.

Exclusion Criteria:

* patient unwillingness to start the procedure without sedation/analgesia
* previous colorectal surgery
* patient refusal or inability to provide informed consent
* inadequate bowel preparation (patients unable to swallow at least ¾ of cleansing preparation, or that did have late and insufficient evacuations, or that reported the presence of residual stools in the last evacuations).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2013-03; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Maximum pain score recorded during colonoscopy. | 1 hour
  Pain will be assessed using a visual analogue scale (VAS) with a score 0=absence of pain, 2=simply "discomfort", 10=the worst possible pain. Before the procedure, an endoscopic nurse will explain the VAS scoring system to the patients. The patient will be informed that the request for pain information is not to remind the patient that the examination should be uncomfortable, but to let the colonoscopist be alerted to the need to use maneuvers to minimize discomfort (e.g. loop reduction, removal of colonic content, abdominal compression and/or change in patient position). At regular intervals during colonoscopy (e.g. every 2-3 minutes) patients will be asked about discomfort or pain. The responses will be recorded, and the maximum pain score noted.

SECONDARY OUTCOMES:
Need for sedation/analgesia and its dosage. | 1 hour
  Sedation and analgesia will be available on demand. Medication will be offered when VAS score reaches ≥2 (discomfort). Patients can accept or decline the medication. If patients agree to accept the medication, it will be given. Midazolam, no more than 5 mg per patient, will be used. When pain is reported, sedation will be started with midazolam with a single intravenous dose of 2 mg, plus incremental doses of 1 mg if the patient still continues to complain about pain. To avoid bias by the colonoscopist, sedation medication will be administered based on the patients' confirmation that the pain is no longer tolerable, and not at the discretion of the colonoscopist. No other analgesic or sedative medications will be administered. The colon segment in which patients requests sedation will be recorded.
Overall pain after the procedure. | 1 hour
  After the procedure and at discharge from the Endoscopy Unit, an assistant nurse blinded to the procedure will ask patients about overall pain using the same VAS when neither the endoscopist nor the assistant nurse who performed the colonoscopy were present. Patients will be asked to quantify the degree of pain experienced and to place a mark over the VAS accordingly.
Cecal intubation rate. | 1 hour
  Cecal intubation will be defined as passage of the tip of the colonoscope beyond the ileocecal valve so that the medial wall of the cecum proximal to the ileocecal valve will be observed. This will be analyzed on an intention- to-treat basis according to group allocation.
Cecal intubation time. | 1 hour
  Cecal intubation time will be defined as the time for passage of the colonoscope from the rectum to the cecum.
Total procedure time. | 1 hour.
  Total procedure time (including time required for polyp resection or biopsy).
Adenoma detection rate. | 10 months.
  Proportion of subjects with at least one adenoma of any size.
Adenoma resection rate. | 10 months.
  Total number of adenomas resected per subject.
Advanced adenoma. | 10 months.
  Total number of advanced adenomas: diameter ≥10mm, or high grade dysplasia, or with ≥20% villous components.

OTHER OUTCOMES:
Position changes. | 1 hour
  Change in patient position as needed if advancement of the colonoscope fails.
Loop reduction maneuvers. | 1 hour
  Applied as needed if advancement of the colonoscope fails.
Amount of water used during the procedure. | 1 hour
  Amount of infused water during insertion and withdrawal.
Bloating at completion of examination. | 1 hour
  Bloating felt by patients at completion of examination on a 10 point visual analogue scale.
Bloating at discharge. | 1 hour
  Bloating felt by patients at discharge measured on a ten point visual analogue scale.
Patients willingness to repeat the examination. | 1 hour
  Patients willingness to repeat the examination based on overall satisfaction about procedure. Measured at discharge on a yes/no question.
Oxygen desaturation. | 1 hour
  Significant oxygen desaturation will be recorded when values less than 85% will be maintained for more than 15 seconds.
Vagal reaction. | 1 hour
  Vagal reaction is defined as heart rate <60 beats per minute accompanied by excessive sweating, nausea and/or vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Cadoni, MD, Principal Investigator — S. Barbara Hospital, Iglesias (CA), Italy
Locations (3):
- Sepulveda Ambulatory Care Center, VA Greater Los Angeles Healthcare System, Los Angeles, California, United States
- Italy (2):
  - S. Barbara Hospital, Iglesias, Cagliari
  - N. S. di Bonaria Hospital, San Gavino Monreale, VS

REFERENCES:
- [Background] Leung FW, Amato A, Ell C, Friedland S, Harker JO, Hsieh YH, Leung JW, Mann SK, Paggi S, Pohl J, Radaelli F, Ramirez FC, Siao-Salera R, Terruzzi V. Water-aided colonoscopy: a systematic review. Gastrointest Endosc. 2012 Sep;76(3):657-66. doi: 10.1016/j.gie.2012.04.467. PMID 22898423
- [Background] Brocchi E, Pezzilli R, Tomassetti P, Campana D, Morselli-Labate AM, Corinaldesi R. Warm water or oil-assisted colonoscopy: toward simpler examinations? Am J Gastroenterol. 2008 Mar;103(3):581-7. doi: 10.1111/j.1572-0241.2007.01693.x. Epub 2007 Dec 12. PMID 18076732
- [Background] Rabenstein T, Radaelli F, Zolk O. Warm water infusion colonoscopy: a review and meta-analysis. Endoscopy. 2012 Oct;44(10):940-51. doi: 10.1055/s-0032-1310157. Epub 2012 Sep 17. PMID 22987214
- [Background] Leung CW, Kaltenbach T, Soetikno R, Wu KK, Leung FW, Friedland S. Water immersion versus standard colonoscopy insertion technique: randomized trial shows promise for minimal sedation. Endoscopy. 2010 Jul;42(7):557-63. doi: 10.1055/s-0029-1244231. Epub 2010 Jun 30. PMID 20593332
- [Background] Leung FW. Water exchange may be superior to water immersion for colonoscopy. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1012-4. doi: 10.1016/j.cgh.2011.09.007. Epub 2011 Sep 22. No abstract available. PMID 21946120
- [Background] Leung F, Harker J, Leung J, Siao-Salera R, Mann S, Ramirez F, Friedland S, Amato A, Radaelli F, Paggi S, Terruzzi V, Hsieh Y. Removal of infused water predominantly during insertion (water exchange) is consistently associated with a greater reduction of pain score - review of randomized controlled trials (RCTs) of water method colonoscopy. J Interv Gastroenterol. 2011 Jul;1(3):114-120. doi: 10.4161/jig.1.3.18510. Epub 2011 Jul 1. PMID 22163081
- [Background] Radaelli F, Paggi S, Amato A, Terruzzi V. Warm water infusion versus air insufflation for unsedated colonoscopy: a randomized, controlled trial. Gastrointest Endosc. 2010 Oct;72(4):701-9. doi: 10.1016/j.gie.2010.06.025. PMID 20883846
- [Background] Pohl J, Messer I, Behrens A, Kaiser G, Mayer G, Ell C. Water infusion for cecal intubation increases patient tolerance, but does not improve intubation of unsedated colonoscopies. Clin Gastroenterol Hepatol. 2011 Dec;9(12):1039-43.e1. doi: 10.1016/j.cgh.2011.06.031. Epub 2011 Jul 13. PMID 21749850
- [Derived] Cadoni S, Sanna S, Gallittu P, Argiolas M, Fanari V, Porcedda ML, Erriu M, Leung FW. A randomized, controlled trial comparing real-time insertion pain during colonoscopy confirmed water exchange to be superior to water immersion in enhancing patient comfort. Gastrointest Endosc. 2015 Mar;81(3):557-66. doi: 10.1016/j.gie.2014.07.029. Epub 2014 Sep 26. PMID 25262100